CLINICAL TRIAL: NCT04552392
Title: Psychological Impact of Institutional Quarantine - A Cross-Sectional Observational Study
Brief Title: Psychological Impact of Institutional Quarantine
Status: Completed | Type: Observational
Sponsor: Dr. Ram Manohar Lohia Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Pragya Sharma, Assistant Professor, Dr. Ram Manohar Lohia Hospital
Other Study IDs: COVID
Record Dates: First submitted 2020-09-15; First posted 2020-09-17 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Quarantine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Quarantine separates persons who have been potentially exposed to an infectious agent (and thus at risk for disease) from the general community. However, it may create psychological, emotional, and financial problems for some persons. The experience of those placed under quarantine in terms of compliance, difficulties, emotional response and psychological impact remains under-researched. In view of the increasing cases of COVID-19 in India and the rising numbers of people being quarantined as a precautionary measure, it was imperative to assess those quarantined for the psychological impact of the concerns regarding this illness and the quarantine procedure. In India, no such study had been undertaken and our study thus filled the research gap. The cross-sectional observational study aims at assessing the psychological impact of quarantine on Indian BSF jawans (n=100). They would be assessed for depression, anxiety, perceived stress level of impact, and impact of life events using Beck Depression Inventory, State Trait Anxiety Inventory, Perceived Stress Scale, and Impact of Events Scale-Revised. A qualitative interview schedule will also be carried out. Data would be analysed.

DETAILED DESCRIPTION:
Institutional quarantine separates persons who have been potentially exposed to an infectious agent (and thus at risk for disease) from the general community. This may create psychological, emotional, and financial problems for some persons. The experience of those placed under quarantine in terms of compliance, difficulties, emotional response and psychological impact remains under-researched.

In view of the increasing cases of COVID-19 in India and the rising numbers of people being quarantined as a precautionary measure, it was imperative to assess those quarantined for the psychological impact of the concerns regarding this illness and the quarantine procedure. In India, no such study had been undertaken and our study would thus fill the research gap.

The cross-sectional observational study is aimed at assessing the psychological impact of quarantine on Indian Border Security Force (BSF) soldiers (n=100).

The participants will be assessed for depression, anxiety, perceived stress level of impact, and impact of life events using Beck Depression Inventory, State Trait Anxiety Inventory, Perceived Stress Scale, and Impact of Events Scale-Revised respectively. A qualitative interview schedule will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Indian-origin adults between the age of 18-60 yrs quarantined at border security force facility
* Both genders would be included

Exclusion Criteria:

* Any chronic co-morbid medical condition
* Current Diagnosis of COVID-19

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Jawana quarantined at Border Security Force Facility as a precautionary measure for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
depression | Baseline
  Beck Depression Inventory
anxiety | Baseline
  State Trait Anxiety Inventory
perceived stress | Baseline
  Perceived Stress Scale
impact of life events | Baseline
  Impact of Events Scale-Revised

CONTACTS AND LOCATIONS:
Overall Officials: Pragya Sharma, PhD, Principal Investigator — Ram Manohar Lohia Hospital
Locations (1):
- ITBP Chawala, Delhi, India

IPD SHARING:
Plan to Share IPD: No